CLINICAL TRIAL: NCT04614571
Title: TCR Sequencing and Transcriptional Profiling in Celiac Disease Patients Undergoing Gluten Challenge
Brief Title: T Cell Receptor (TCR) Sequencing and Transcriptional Profiling in Adult Celiac Disease Patients Undergoing Gluten Challenge
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0000-CD-CES-1880
Record Dates: First submitted 2020-09-24; First posted 2020-11-04 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Celiac Disease
Keywords: CeD; HLA-DQ2 positive; HLA-DQ8 positive
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gluten Challenge (Other)
  Interventions: Dietary Supplement: Gluten Powder

INTERVENTIONS:
Dietary Supplement: Gluten Powder — Administered orally daily for 14 days

SUMMARY:
The primary objectives are:

* Characterize the T cell receptor (TCR) repertoire in duodenal biopsy samples of participants pre- and post-challenge.
* Compare for each patient the TCR repertoire of duodenal biopsy samples with the peripheral blood TCR repertoire of each study participant
* Characterize the transcriptome of duodenal biopsy samples and blood from study participants pre- and post-challenge

The secondary objectives are:

* Ex vivo identification and validation of DQ-restricted gliadin specific TCRs.
* Characterize the gluten-challenge induced changes in small intestine histology using standard for Celiac Disease (CeD) histological assessments

ELIGIBILITY:
Key Inclusion Criteria:

1. Have a body mass index (BMI) ≥17 and ≤40 kg/m2 and a body weight >45 kg at the Screening Visit
2. Be judged to be in good health as defined in the protocol
3. Have well-controlled biopsy-proven CeD, compliant with a GFD for ≥6 months preceding Screening as defined in the protocol
4. Be HLA-DQ2 and/or HLA-DQ8 positive as defined in the protocol

Key Exclusion Criteria:

1. Have a history of gluten triggered acute symptoms (≤24 hours after gluten exposure), and/or severe symptoms (abdominal pain interfering with daily activities, diarrhea with >5 stools/day), and/or prolonged symptoms (duration >7 days)
2. Have a history of clinically significant endocrine, cardiovascular, hematological, hepatic, immunological (other than CeD or autoimmune thyroid disease), renal, respiratory, genitourinary, or major neurological (including stroke and chronic seizures) abnormalities or disease
3. Have participated in another investigational trial within 4 weeks before Screening
4. Have a history of cancer (malignancy) other than nonmelanoma skin cancer
5. Have a history of significant multiple and/or severe allergies (e.g., latex allergy)
6. Presence of HIV (HIV Ab), hepatitis B (HBsAg, HBAb) or Hepatitis C (HCV Ab) seropositivity at screening
7. Ongoing immunosuppression or receive any treatment that might alter T cell repertoire or phenotype

Note: Other protocol-defined inclusion/ exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-11-02 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in small intestine TCR repertoire | Up to 30 days post challenge
  Change in the T-cell receptor repertoire (measured by T cell receptor sequencing) in the small intestine after gluten challenge
Change from Baseline in peripheral blood TCR repertoire | Up to 30 days post challenge
  Change in the T-cell receptor repertoire (measured by T cell receptor sequencing) in peripheral blood after gluten challenge
Changes from baseline in small intestine and peripheral blood transcriptome | Up to 30 days post challenge
  Change in the gene expression profile (transcriptomic analysis by ribonucleic acid [RNA] sequencing and cellular indexing of transcriptomes and epitopes by sequencing [CITEseq]) of the small intestine and peripheral blood after gluten challenge

SECONDARY OUTCOMES:
Change from Baseline in Small Intestine Histology Based on Intraepithelial Lymphocytes (IEL) Count per 100 epithelial cells | Baseline and Day 15
  IELs are white blood cells (WBCs) interspersed between epithelial cells of the small and large intestine where they function to preserve the integrity of the mucosal barrier by protecting the epithelium against pathogen or immune-induced pathology. Increased IELs count indicated more extreme CeD disease symptoms. Baseline values are defined as the last observed value before the first dose of gluten.
Change from Baseline in Small Intestine Histology Based on Villous Height (Microns), Crypt Depth (Microns) and Villous Height to Crypt Depth Ratio (Vh:Cd) | Baseline and Day 15
  Villi are the small finger like projections that line the small intestine and promote nutrient absorption and are often shortened in active CeD. Crypts are grooves between the villi that are often elongated in CeD. A decreased Vh:Cd ratio indicates more extreme CeD disease symptoms. Baseline values (Microns) will be defined as the last observed value before the first dose of gluten.
Identification and ex vivo functional validation of gluten-specific T cells | Up to 30 days post challenge
  Clonality of peripheral blood mononuclear cell (PBMC)-derived gluten-specific T cells (measured by T cell receptor sequencing) after ex vivo expansion with gluten peptides

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Administrator, Study Director — Regeneron Pharmaceuticals
Locations (1):
- Celiac Research Centre Mass General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/